CLINICAL TRIAL: NCT05766449
Title: Risk Factors for Hepatic Inflammation, Fibrosis and Prognosis in Patients With Chronic Hepatitis B Combined With Non-alcoholic Fatty Liver Disease
Brief Title: Risk Factors for Hepatic Inflammation, Fibrosis and Prognosis in Patients With CHB and NAFLD
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jie Li, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: CHB AND NAFLD
Record Dates: First submitted 2023-02-21; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Chronic Hepatitis b; Non-alcoholic Fatty Liver Disease
Keywords: chronic hepatitis b; nonalcoholic fatty liver diabetes; inflammation; fibrosis; prognosis
MeSH Terms: conditions — Hepatitis B, Chronic; Non-alcoholic Fatty Liver Disease; Inflammation; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic hepatitis B (CHB) affects an estimated 292 million people, and causes approximately 800,000 people deaths per year from liver-related complications including cirrhosis and hepatocellular carcinoma, remaining a major global public health issue.Meanwhile, with the improvement of living standards and changes in lifestyle and dietary habits, non-alcoholic fatty liver disease (NAFLD) has become another important cause of liver cirrhosis and HCC.HBV combined with NAFLD inevitably develops into continuous or intermittent liver inflammation and fibrosis, which greatly increases the risk of cirrhosis, liver cancer and even end-stage liver disease. We aimed to investigate the risk factors and establish diagnostic models for hepatic inflammation, fibrosis in patients with CHB associated NAFLD. In addition, to find risk factors for liver cirrhosis, liver cancer or liver failure in patients with CHB-related NAFLD.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) affects an estimated 292 million people, and causes approximately 800,000 people deaths per year from liver-related complications including cirrhosis and hepatocellular carcinoma, remaining a major global public health issue.Meanwhile, with the improvement of living standards and changes in lifestyle and dietary habits, non-alcoholic fatty liver disease (NAFLD) has become another important cause of liver cirrhosis and HCC.HBV combined with NAFLD inevitably develops into continuous or intermittent liver inflammation and fibrosis, which greatly increases the risk of cirrhosis, liver cancer and even end-stage liver disease. We aimed to investigate the risk factors and establish diagnostic models of hepatic inflammation and fibrosis in CHB associated NAFLD patients using a multicenter study. In addition, to find risk factors for liver cirrhosis, liver cancer or liver failure in patients with CHB-related NAFLD.

ELIGIBILITY:
Inclusion Criteria:

1.18 years or older 2. Positive hepatitis B surface antigen (HBsAg) for at least 6 months and without other viral co-infection at baseline 2.NAFLD diagnosed by imaging liver biopsy, and/or blood testing/predictive indices

Exclusion Criteria:

1. Other chronic liver diseases, such as alcoholic liver disease, other viral hepatitis, drug-induced liver injury;
2. HCC or other malignancies before liver biopsy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic hepatitis B (CHB) patients concurrent with nonalcoholic fatty liver disease (NAFLD)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Risk factors for hepatic inflammation or fibrosis in chronic hepatitis B patients with non-alcoholic fatty liver disease | 0 year
  Risk factors for hepatic inflammation or fibrosis in patients with chronic hepatitis B and non-alcoholic fatty liver disease at baseline
Risk factors of chronic hepatitis B patients with non-alcoholic fatty liver disease progressing to cirrhosis, liver cancer or liver failure | 1 year
  Risk factors of chronic hepatitis B patients with non-alcoholic fatty liver disease progressing to cirrhosis, liver cancer or liver failure during 1-year follow-up
Risk factors of chronic hepatitis B patients with non-alcoholic fatty liver disease progressing to cirrhosis, liver cancer or liver failure | 3 years
  Risk factors of chronic hepatitis B patients with non-alcoholic fatty liver disease progressing to cirrhosis, liver cancer or liver failure during 3-year follow-up
Risk factors of chronic hepatitis B patients with non-alcoholic fatty liver disease progressing to cirrhosis, liver cancer or liver failure | 5 years
  Risk factors of chronic hepatitis B patients with non-alcoholic fatty liver disease progressing to cirrhosis, liver cancer or liver failure during 5-year follow-up

SECONDARY OUTCOMES:
Establishment a diagnostic model for hepatic inflammation in chronic hepatitis B patients with non-alcoholic fatty liver disease | 0 year
  Establishment a diagnostic model of hepatic inflammation in chronic hepatitis B patients with non-alcoholic fatty liver disease using baseline data
Establishment a diagnostic model for hepatic fibrosis in patients with chronic hepatitis B and non-alcoholic fatty liver disease | 0 year
  Establishment a diagnostic model for hepatic fibrosis in chronic hepatitis B patients with non-alcoholic fatty liver disease using baseline data
Establishment predictive models for the progression of chronic hepatitis B patients with non-alcoholic fatty liver disease to cirrhosis, liver cancer or liver failure | 1 year
  Establishment predictive models for the progression of chronic hepatitis B patients with non-alcoholic fatty liver disease to cirrhosis, liver cancer or liver failure within one year
Establishment predictive models for the progression of chronic hepatitis B patients with non-alcoholic fatty liver disease to cirrhosis, liver cancer or liver failure | 3 years
  Establishment predictive models for the progression of chronic hepatitis B patients with non-alcoholic fatty liver disease to cirrhosis, liver cancer or liver failure within 3 years
Establishment predictive models for the progression of chronic hepatitis B patients with non-alcoholic fatty liver disease to cirrhosis, liver cancer or liver failure | 5 years
  Establishment predictive models for the progression of chronic hepatitis B patients with non-alcoholic fatty liver disease to cirrhosis, liver cancer or liver failure within 5 years
Incidence of cirrhosis, cancer and liver failure in patients with chronic hepatitis B and non-alcoholic fatty liver disease | 5 years
  Incidence of cirrhosis, cancer and liver failure in patients with chronic hepatitis B and non-alcoholic fatty liver disease for 1 year, 3 years and 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, China

REFERENCES:
- [Derived] Rui F, Xu L, Yeo YH, Xu Y, Ni W, Tan Y, Zheng Q, Tian X, Zeng QL, He Z, Qiu Y, Zhu C, Ding W, Wang J, Huang R, Xue Q, Wang X, Chen Y, Fan J, Fan Z, Ogawa E, Kwak MS, Qi X, Shi J, Wong VW, Wu C, Li J. Machine Learning-Based Models for Advanced Fibrosis and Cirrhosis Diagnosis in Chronic Hepatitis B Patients With Hepatic Steatosis. Clin Gastroenterol Hepatol. 2024 Nov;22(11):2250-2260.e12. doi: 10.1016/j.cgh.2024.06.014. Epub 2024 Jun 19. PMID 38906440
- [Derived] Rui F, Yeo YH, Xu L, Zheng Q, Xu X, Ni W, Tan Y, Zeng QL, He Z, Tian X, Xue Q, Qiu Y, Zhu C, Ding W, Wang J, Huang R, Xu Y, Chen Y, Fan J, Fan Z, Qi X, Huang DQ, Xie Q, Shi J, Wu C, Li J. Development of a machine learning-based model to predict hepatic inflammation in chronic hepatitis B patients with concurrent hepatic steatosis: a cohort study. EClinicalMedicine. 2024 Jan 16;68:102419. doi: 10.1016/j.eclinm.2023.102419. eCollection 2024 Feb. PMID 38292041